CLINICAL TRIAL: NCT04530396
Title: Randomized Double-blind Placebo-controlled Multi-center Clinical Trial in Parallel Assignment of Efficacy, Safety, and Immunogenicity of Gam-COVID-Vac Combined Vector Vaccine in SARS-СoV-2 Infection Prophylactic Treatment
Brief Title: Clinical Trial of Efficacy, Safety, and Immunogenicity of Gam-COVID-Vac Vaccine Against COVID-19
Acronym: RESIST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Government of the city of Moscow (Unknown); CRO: Crocus Medical BV (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-Gam-COVID-Vac-2020
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-08

CONDITIONS: Covid19 Prevention
Keywords: COVID-19; vector vaccine; SARS-CoV-2; adenoviral vector
MeSH Terms: conditions — COVID-19 | interventions — Gam-COVID-Vac vaccine

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Group (Experimental): Gam-COVID-Vac combined vector vaccine, 0,5ml/dose+0,5 ml/dose prime-boost immunization in days 1 (component I rAd26-S) and 21(component II rAd5-S)
  Interventions: Biological: Gam-COVID-Vac
- Control Group (Placebo Comparator): placebo, 0,5ml/dose+0,5 ml/dose immunization in days 1 and 21
  Interventions: Other: placebo

INTERVENTIONS:
Biological: Gam-COVID-Vac — vaccine for intramuscular injection
  Arms: Primary Group
Other: placebo — placebo comparator
  Arms: Control Group

SUMMARY:
Randomized, double-blind (blinded for the trial subject and the study physician), placebo controlled, multi-center clinical trial in parallel assignment of efficacy, immunogenicity, and safety of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection in adults in the SARS-СoV-2 infection prophylactic treatment.

DETAILED DESCRIPTION:
Randomized, double-blind (blinded for the trial subject and the study physician), placebo controlled, multi-center clinical trial in parallel assignment of efficacy, immunogenicity, and safety of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection in adults in the SARS-СoV-2 infection prophylactic treatment.

The trial will include 40,000 volunteers aged 18+. After screening, they will be randomized (3:1) into two groups - a reference group of 10,000 volunteers receiving placebo and a study group of 30,000 volunteers receiving the Gam-COVID-Vac combined vector vaccine against the SARS-СoV-2-induced coronavirus infection.

The trial subjects will be randomized into five age strata: 18-30, 31-40, 41-50, 51-60, and 60+ years.

The PCR test for SARS-CoV-2 RNA detection at the visit is performed during screening and before the second administration of the vaccine/placebo

Each subject will participate in the trial for 180±14 days after the first dose of the study drug/placebo and will have one screening visit and five on-site visits to the study physician during the said period. The study drug/placebo will be administered intramuscularly during vaccination visits 1 and 2 (day 0 and day 21±2). Subsequent observation visits 3, 4, and 5 will be made on days14±2, 28±2, 35±2,42±2, and 180±14 respectively. During the observation visits, vital signs will be assessed in all trial subjects and changes in the subjects' condition and wellbeing compared to the previous visit will be recorded. Observation visits may be remote, through the telemedicine consultation (TMC).

Additionally, the trial subjects will be able to have remote consultations with the physician through the TMC.

Blood samples will be taken from certain subjects during the following visits to assess the immunogenicity parameters listed below:

Virus-neutralizing activity (300 subjects) ×3 Interferon gamma (107 subjects) ×3 CD4 and CD8 cell count and ratio (50 subjects) SARS-CoV-2 glycoprotein-specific antibodies titer (9,520 subjects) ×3 Determination of the titer of SARS-CoV-2 nucleocleocapsid protein-specific antibodies(9,520 subjects) ×3

Blood sampling will be performed on the day of injecting the first dose of the study drug/placebo immediately prior to the study drug administration Blood sampling for immunogenicity parameters assessment will be only carried out in specially selected study centers.

Blood samples will be taken from 9,520 trial subjects. All four immunogenicity parameters may be assessed in one trial subject.

Trial subjects data will be collected using electronic case report forms and electronic questionnaires to be filled by trial subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of a subject to participate in the trial
2. Males and females aged ≥18 y.o.;
3. Negative HIV, hepatitis, and syphilis test results
4. Negative anti-SARS CoV2 IgM and IgG antibodies test carried out with the enzyme immunoassay method
5. Negative COVID-2019 PCR test result at the screening visit
6. No COVID-2019 in the past medical history
7. No contact with COVID-2019 diseased persons within at least 14 days before the enrollment (according to trial subjects)
8. Consent to use effective contraception methods during the trial
9. Negative urine pregnancy test at the screening visit (for child-bearing age women)
10. Negative drugs or psychostimulants urine test at the screening visit
11. Negative alcohol test at the screening visit
12. No evident vaccine-induced reactions or complications after receiving immunobiological products in the past medical history
13. No acute infectious and/or respiratory diseases within at least 14 days before the enrollment.

Exclusion Criteria:

1. Any vaccination/immunization within 30 days before the enrollment;
2. Steroids (except hormonal contraceptives) and/or immunoglobulins or other blood products therapy not finished 30 days before the enrollment
3. Immunosuppressors therapy finished within 3 months before the enrollment
4. Pregnancy or breast-feeding
5. Acute coronary syndrome or stroke suffered less than one year before the enrollment
6. Tuberculosis, chronic systemic infections
7. Drug allergy (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, atopy, serum disease), hypersensitivity or allergic reaction to immunobiological products, known allergic reactions to study drug components, acute exacerbation of allergic diseases on the enrollment day
8. Neoplasms in the past medical history (ICD codes C00-D09)
9. Donated blood or plasma (450+ ml) within 2 months before the enrollment
10. History of splenectomy;
11. Neutropenia (absolute neutrophil count <1,000/mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin <80 g/L), immunodeficiency in the past medical history within 6 months before the enrollment
12. Active form of a disease caused by the human immunodeficiency virus, syphilis, hepatitis B or C
13. Anorexia, protein deficiency of any origin
14. Big-size tattoos at the injection site (deltoid muscle area), which does not allow assessing the local response to the study drug/placebo administration
15. Alcohol or drug addiction in the past medical history
16. Participation in any other interventional clinical trial
17. Any other condition that the study physician considers as a barrier to the trial completion as per the protocol
18. Study center staff or other employees directly involved in the trial, or their families.

If a subject has any contraindications to vaccination based on the Guidelines on Detection, Investigation and Prevention, of Vaccination-induced Side Reactions (approved by the Ministry of Healthcare of Russia on Apr. 12, 2019, the vaccination may be postponed for a period of time specified in the document.

Ages: 18 Years to 111 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33758 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
percentage of trial subjects with coronavirus disease 2019 (COVID-19) developed within 6 months after the first dose | through the whole study, an average of 180 days
  Demonstrate the superiority of Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection compared to placebo, based on the percentage of trial subjects with coronavirus disease 2019 (COVID-19) developed within 6 months after the second dose of the study drug/placebo, as confirmed with the method of polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
the severity of the clinical course of COVID-19 | through the whole study, an average of 180 days
  Assess the efficacy of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus compared to placebo, based on the severity of the clinical course of COVID-19
Changing of antibody levels against the SARS-CoV-2 glycoprotein S | day before injecting the first dose of the study drug/placebo and 42±2 and 180±14 days after the first dose
  Assess the immunogenicity of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection compared to placebo, based on the geometric mean titer of SARS-CoV-2 glycoprotein-specific antibodies
Changing of antigen-specific cellular immunity level | the drug administration day before injecting the first dose of the study drug/placebo and 28±2 days after the first dose
  Describe the strength of cell-mediated immune response induced by the use of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection compared to placebo
Changing of of virus neutralizing antibody titer | the drug administration day before injecting the first dose of the study drug/placebo and 42±2 days after the first dose
  Geometric mean virus-neutralizing antibodies titer
Incidence of adverse events in trial subjects | through the whole study, an average of 180 days
  Incidence of adverse events in trial subjects compared to placebo
Severity of adverse events in trial subjects | through the whole study, an average of 180 days
  Severity of adverse events in trial subjects compared to placebo
estimation of the proportion of study subjects with antibodies to the N-protein of the virus SARS-CoV-2 | day before injecting the first dose of the study drug/placebo and 42±2 and 180±14 days after the first dose
  Percentage of study subjects with antibodies
  to the N-protein of the SARS - CoV-2 virus that appeared after
  vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Elena Smolyarchuk, MD, PhD, Study Chair — Study Coordinator; Sergey Zyryanov, MD, PhD, Study Chair — Study Coordinator
Locations (23):
- Russia (23):
  - ARCHIMED V Clinic of new medical technologies limited liability company, Moscow
  - Hadassah LTD, Moscow
  - Medsi Group of companies joint-stock company", Moscow
  - Niarmedic Plus, Moscow
  - State budgetary healthcare institution of the city of Moscow "City clinical hospital No. 52 of the Moscow city health Department", Moscow
  - State Budgetary Healthcare Institution, Moscow, Consultation and Diagnosis Polyclinic No. 121, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, M. Konchalovsky Municipal Clinical Hospital, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, M. Zhadkevich Municipal Clinical Hospital, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 115, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 2, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 210, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 212, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 219, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Moscow, Municipal Polyclinic No. 220, Moscow Healthcare Department, Moscow
  - State Budgetary Healthcare Institution, Municipal Polyclinic No. 62, Moscow Healthcare Department, Moscow
  - State budgetary institution of health care of the city of Moscow " city polyclinic No. 109 Of the Department of health of the city of Moscow", Moscow
  - State budgetary institution of health care of the city of Moscow " city polyclinic No. 170 Of the Department of health of the city of Moscow", Moscow
  - State budgetary institution of health care of the city of Moscow " city polyclinic No. 36 Of the Department of health of the city of Moscow", Moscow
  - State budgetary institution of health care of the city of Moscow " city polyclinic No. 46 Of the Department of health of the city of Moscow", Moscow
  - State budgetary institution of health care of the city of Moscow " city polyclinic No. 6 Of the Department of health of the city of Moscow", Moscow
  - State budgetary institution of health care of the city of Moscow " city polyclinic No. 68 Of the Department of health of the city of Moscow", Moscow
  - State budgetary institution of health care of the city of Moscow "Diagnostic center No. 5 with polyclinic Department Of the Department of health of the city of Moscow", Moscow
  - State budgetary institution of health care of the city of Moscow "Diagnostic clinical center No. 1 Of the Department of health of the city of Moscow", Moscow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Logunov DY, Dolzhikova IV, Shcheblyakov DV, Tukhvatulin AI, Zubkova OV, Dzharullaeva AS, Kovyrshina AV, Lubenets NL, Grousova DM, Erokhova AS, Botikov AG, Izhaeva FM, Popova O, Ozharovskaya TA, Esmagambetov IB, Favorskaya IA, Zrelkin DI, Voronina DV, Shcherbinin DN, Semikhin AS, Simakova YV, Tokarskaya EA, Egorova DA, Shmarov MM, Nikitenko NA, Gushchin VA, Smolyarchuk EA, Zyryanov SK, Borisevich SV, Naroditsky BS, Gintsburg AL; Gam-COVID-Vac Vaccine Trial Group. Safety and efficacy of an rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine: an interim analysis of a randomised controlled phase 3 trial in Russia. Lancet. 2021 Feb 20;397(10275):671-681. doi: 10.1016/S0140-6736(21)00234-8. Epub 2021 Feb 2. PMID 33545094